CLINICAL TRIAL: NCT02022163
Title: Safety, Tolerability and Immunogenicity of a Plant-made H7 Virus-like Particle (VLP) Influenza Vaccine in Adults.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medicago (Industry)
Collaborators: Health Sciences Centre, Winnipeg, Manitoba (Other); Public Health Agency of Canada (PHAC) (Other Government); Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CP-H7VLP-006
Record Dates: First submitted 2013-12-20; First posted 2013-12-27 (Estimated); Last update posted 2015-09-25 (Estimated); Status verified 2015-09

CONDITIONS: Virus Diseases; RNA Virus Infections; Respiratory Tract Diseases; Respiratory Tract Infections
Keywords: Influenza, Human; RNA Virus Infections; Respiratory Tract Diseases; Respiratory Tract Infections; Aluminum Hydroxide; Adjuvants, Immunologic; Immunogenic Factors; Physiological Effects of Drugs; Virus Diseases; Orthomyxoviridae Infections; Infection
MeSH Terms: conditions — Virus Diseases; RNA Virus Infections; Respiratory Tract Diseases; Respiratory Tract Infections; Influenza, Human; Orthomyxoviridae Infections; Infections | interventions — Aluminum Hydroxide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Low dose of H7 VLP vaccine + Alhydrogel (Experimental): Biological: Low dose of H7 VLP vaccine mixed with Alhydrogel, 2 doses given 21 days apart
  Interventions: Biological: Low dose of H7 VLP vaccine + Alhydrogel
- Med dose of H7 VLP vaccine + Alhydrogel (Experimental): Biological: Med dose of H7 VLP vaccine mixed with Alhydrogel, 2 doses given 21 days apart
  Interventions: Biological: Med dose of H7 VLP vaccine + Alhydrogel
- High dose of H7 VLP vaccine + Alhydrogel (Experimental): Biological: High dose of H7 VLP vaccine mixed with Alhydrogel, 2 doses given 21 days apart
  Interventions: Biological: High dose of H7 VLP vaccine + Alhydrogel
- High dose of H7 VLP vaccine (Experimental): Biological: High dose of H7 VLP vaccine, 2 doses given 21 days apart
  Interventions: Biological: High dose of H7 VLP vaccine
- Placebo (Placebo Comparator): Placebo, 2 doses given 21 days apart
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Low dose of H7 VLP vaccine + Alhydrogel — Low dose of H7 VLP vaccine mixed with Alhydrogel, 2 doses given 21 days apart
  Arms: Low dose of H7 VLP vaccine + Alhydrogel
Biological: Med dose of H7 VLP vaccine + Alhydrogel — Med dose of H7 VLP vaccine mixed with Alhydrogel, 2 doses given 21 days apart
  Arms: Med dose of H7 VLP vaccine + Alhydrogel
Biological: High dose of H7 VLP vaccine + Alhydrogel — High dose of H7 VLP vaccine mixed with Alhydrogel, 2 doses given 21 days apart
  Arms: High dose of H7 VLP vaccine + Alhydrogel
Biological: High dose of H7 VLP vaccine — High dose of H7 VLP vaccine, 2 doses given 21 days apart
  Arms: High dose of H7 VLP vaccine
Biological: Placebo — Placebo, 2 doses given 21 days apart
  Arms: Placebo

SUMMARY:
A phase I trial conducted in a single centre, observer-blind, randomized, dose-ranging, placebo-controlled study to evaluate the safety, tolerability, and immunogenicity of 2 intramuscular injections of plant-based H7 VLP Influenza Vaccine administered to healthy adults, 18-60 years of age.

DETAILED DESCRIPTION:
This study will consist of a dose-ranging in one hundred (100) subjects who will be randomized in parallel to a 1:1:1:1:1 ratio in five (5) groups of 20 subjects to receive one intramuscular injection at Days 0 and 21 of either a low, medium or high dose of H7 VLP vaccine mixed with Alhydrogel® 0.4% (0.5 mg Aluminum per dose) or a high dose of H7 VLP alone or the placebo preparation (100 millimolar (mM) phosphate buffer + 150 mM sodium chloride (NaCl) + 0.01% Tween 80). Twenty-one (21) days after each immunization, key safety and immunogenicity data will be collected and analysed. All subjects will be followed for safety until Day 228.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults, 18 to 60 years of age, inclusive
* Healthy as judged by the Investigator or designee and determined by medical history, complete general history/symptom-directed physical examination, vital signs, screening laboratories, and medical history conducted no more than 30 days prior to study vaccine administration
* BMI of ≥18 and ≤32
* Comprehension of the study requirements, expressed availability for the required study period, and ability to attend scheduled visits
* Accessible by phone on a consistent basis
* Give his/her consent to participate in this study (by signing the ICF). In the opinion of the Investigator, competence and willingness to provide written, informed consent for participation after reading the informed consent form. The subject must have adequate opportunity to discuss the study with an Investigator or qualified designee
* If female, have a negative pregnancy test result prior to first immunization
* Female of childbearing potential (except subjects in a monogamous same sex relationship), must use an effective birth control for the 28 days prior to immunization and must agree to continue employing adequate birth control measures from Day 0 (first immunization) until at least 60 days post-second immunization and must have no plan to become pregnant from Day 0 (first immunization) until at least 60 days post-second immunization. Highly effective birth control includes hormonal contraceptives (e.g., injectable, topical [patch], estrogenic vaginal ring, etc.), intra-uterine device (IUD), abstinence (confirmed by Investigator), or male condom plus spermicide. Abstinent subjects should be asked what method(s) they would use, should their circumstances change, and subjects without a well-defined plan should be excluded

Exclusion Criteria:

* Presence of significant acute or chronic, uncontrolled medical or neuropsychiatric illness. "Uncontrolled" is defined as
* Requiring a new medical or surgical treatment within one month prior to study vaccine administration
* Requiring a change in medication dosage in one month prior to study vaccine administration due to uncontrolled symptoms or drug toxicity (elective dosage adjustments in stable subjects are acceptable)
* Hospitalization or an event fulfilling the definition of a serious adverse event within one month prior to study vaccine administration
* Any medical or neuropsychiatric condition or any history of excessive alcohol use or drug abuse which, in the Investigator's opinion, would render the subject incompetent to provide informed consent or unable to provide valid safety observations and reporting
* Any confirmed or suspected immunosuppressive condition or immunodeficiency including history of human immunodeficiency virus (HIV) infection, Hepatitis B or C, or the presence of lymphoproliferative disease
* Presence of any febrile illness, oral temperature of >38.0˚C within 24 hours prior to immunization. Such subjects may be re-evaluated for enrolment after resolution of illness
* History of autoimmune disease
* Administration of any vaccine (including any other influenza vaccine) within 30 days prior to study enrolment or planned administration within the period from the vaccination up to blood sampling at Day 42 or within 30 days prior to blood sampling at Day 228. Immunization on an emergency basis of a tetanus and diphtheria toxoids adsorbed for adult use (Td) will be allowed provided the vaccine is not administered within two weeks prior to study vaccine administration. Receipt of any other emergency immunizations (e.g., rabies) will result in a case-by-case review by the medical monitor of continued participation
* Administration of any adjuvanted or investigational influenza vaccine other than a 'simple' seasonal Trivalent Inactivated Vaccine (TIV) or Quadrivalent Inactivated Vaccine (QIV) within 1 year prior to study enrolment or planned administration prior to the end of this trial (Day 228)
* Use of any investigational or non-registered product within 30 days prior to study enrolment or planned use during the study period. Subjects may not participate in any other investigational or marketed drug study while participating in this study
* Treatment with systemic glucocorticoids at a dose exceeding 10 mg of prednisone per day, or equivalent for more than 7 consecutive days or for 10 or more days in total, within one month of study vaccine administration, any other cytotoxic or immunosuppressant drug, or any globulin preparation within 3 months of vaccination. Low doses of nasal or inhaled glucocorticoids are generally allowed
* Use of high dose inhaled steroids or oral and parenteral high dose steroid medications. Nasal steroids are allowed
* Any significant disorder of coagulation or treatment with warfarin derivatives or heparin. Persons receiving prophylactic anti-platelet medications, e.g., low-dose aspirin [≤ 325 mg/day (1 regular adult aspirin) or ≤ 81 mg/day (1 baby aspirin)], and without a clinically apparent bleeding tendency are eligible
* History of previous H7N9 vaccination or a history of exposure to H7N9 virus. Any subject that was enrolled on previous H7N9 studies (except the ones that received placebo) would not be eligible
* Are at high risk of contracting H7N9 influenza infection (e.g. poultry workers)
* History of allergy to any of the constituents of the H7 VLP (H7N9) study vaccine, Alhydrogel® (aluminum hydroxide), or to the phosphate-buffered saline (PBS) (used as placebo)
* History of severe allergic reactions (including anaphylaxis) to any food, medication or bee sting or previous severe asthma.
* History of tobacco allergy
* Continuous use of anti-histamines in the last 4 weeks prior to first immunization or use of anti-histamines 48 hours prior to each study immunization
* Have a rash, dermatological condition, tattoos, or muscle mass at injection site which may interfere with injection site reaction rating
* Have received a blood transfusion within 90 days prior to study vaccination
* If female, positive pregnancy test results at screening, and prior to immunizations on Day 0 and Day 21
* Female subjects who are lactating
* Any vital sign abnormalities: systolic blood pressure, diastolic blood pressure, resting heart rate not well controlled or according to the Investigator's opinion
* Cancer or treatment for cancer within 3 years of study vaccine administration. Persons with a history of cancer who are disease-free without treatment for 3 years or more are eligible. Persons with treated and uncomplicated basal cell carcinoma of the skin are eligible

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2013-12; Primary Completion 2014-09 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Safety | 21 days after each injection and 6-month follow-up period
  Safety will be assessed by the rate, severity and relationship to vaccination of solicited and unsolicited adverse events post-vaccinations. A 6-month follow-up period will be performed.
Immunogenicity | 21 days after each injection
  Geometric mean titers (GMTs) of hemagglutination inhibition (HI antibody on Days 0, 21 and 42 to measure Geometric mean fold rise (GMFR) and seroconversion rates).

SECONDARY OUTCOMES:
Immunogenicity 2 | 21 days after injection and 6-month follow up
  Geometric mean titers (GMTs) of hemagglutination inhibition (HI antibody on Days 0, 21 and 42 to measure seroprotection rates). Follow-up serology samples for GMTs will be taken at Day 228.
Immunogenicity 3 | 21 days after each injection and 6 months follow up
  Geometric mean titers (GMTs) of hemagglutination inhibition against heterologous influenza strains for cross-reactivity assessment. HI antibody on Days 0, 21 and 42 to measure seroconversion rates, GMFR and seroprotection rates. Follow-up serology samples for GMTs will be taken at Day 228.

CONTACTS AND LOCATIONS:
Overall Officials: Neil Simonsen, MD, Principal Investigator — Canadian Science Centre for Human and Animal Health
Locations (1):
- Canadian Science Centre for Human and Animal Health, Winnipeg, Manitoba, Canada